CLINICAL TRIAL: NCT01634178
Title: A Phase 1, Open-Label, Randomized, Two-Period, Two-Sequence Crossover Study to Assess the Effect of Food on the Pharmacokinetics of a Single 30 mg Tablet of Apremilast (CC-10004) in Healthy Subjects
Brief Title: Effect of Food on the Pharmacokinetics of Apremilast (CC-10004) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-CP-022; 20200148 (Other: Amgen Study ID)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteer
Keywords: Apremilast,; pharmacokinetic; safety; Safety and pharmacokinetics in healthy volunteer subjects
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: Apremilast Fasted / Fed (Experimental): In Period 1 participants will receive a single 30 mg apremilast tablet administered under fasted conditions and in Period 2 participants will receive a single 30 mg apremilast tablet administered after a high fat meal.
  Interventions: Drug: Apremilast
- Sequence 2: Apremilast Fed / Fasted (Experimental): In Period 1 participants will receive a single 30 mg apremilast tablet administered after a high fat meal and in Period 2 participants will receive a single 30 mg apremilast tablet administered under fasted conditions.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Tablet for oral administration
  Other Names: CC-10004; Otezla®

SUMMARY:
The purpose of the study is to evaluate the effects of a high fat meal on the pharmacokinetics of a single dose of 30 mg apremilast in healthy adults.

DETAILED DESCRIPTION:
Participants will be randomized to receive a single dose of 30 mg apremilast during each of the 2 periods; once under fasting conditions and once after a high fat meal. Participants will be randomly assigned to receive apremilast either fasted first, then fed, or fed first then fasted. Participants will check into the study center on Day -1 of each period, will be dosed on Day 1, and discharged from the study center on Day 3 after all scheduled pharmacokinetic blood draws and safety evaluations. After a washout of 5 to 10 days, participants will return for period 2 during which they will receive apremilast according to their assigned sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects of any ethnic origin between ages of 18 and 65 inclusive with a body mass index (BMI) between 18 and 33.
2. Females who are able to become pregnant have a negative pregnancy test at screening and baseline, and must agree to use one of the following:

   * a highly effective form of contraception (ex. Non-oral hormonal, intrauterine device) OR
   * oral hormonal contraceptive plus one additional form of barrier contraception OR
   * Two forms of barrier contraception These must be effective by the time of screening.
3. All other females must have been surgically sterilized at least 6 months prior to screening or be postmenopausal (to be confirmed by lab tests).
4. Males must agree to use latex or polyurethane condoms when engaging in sex during the study and for at least 28 days after dosing.

Exclusion Criteria:

1. Any condition, including the presence of laboratory abnormalities, or psychiatric illness, that would prevent the subject from signing the Informed Consent form, places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
2. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, or plans to have elective or medical procedures during the conduct of the trial.
3. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
4. Subjects with known serum hepatitis, is a known carrier of hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus antibody.
5. Subjects who have used prescription systemic or topical medications within 30 days of dosing, unless it is being used to treat a stable, chronic medical condition. This includes medication that is an inhibitor or inducer of P-glycoprotein transporter and CYP-3A4/5 used within 14 days of dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- PPD Development, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinical research site in the United States.
Pre-assignment Details: The study consisted of 2 periods. Participants were randomly assigned to one of two treatment sequences; Fasted then Fed or Fed then Fasted. Each participant was to receive 1 dose of apremilast under fasted conditions and 1 dose of apremilast under fed conditions in each period, respectively, depending on their sequence assignment.
  There was a 5 to 10 day washout period between each dose.
Groups:
- Sequence 1: Apremilast Fasted / Fed: Participants were randomized to receive a single 30 mg apremilast tablet administered under fasted conditions in Period 1 and a single 30 mg apremilast tablet administered after a high fat meal in Period 2.
- Sequence 2: Apremilast Fed / Fasted: Participants were randomized to receive a single 30 mg apremilast tablet administered after a high fat meal in Period 1 and a single 30 mg apremilast tablet administered under fasted conditions in Period 2.
Period: Treatment Period 1
Arm/Group | Sequence 1: Apremilast Fasted / Fed | Sequence 2: Apremilast Fed / Fasted
Started | 23 | 23
Completed | 23 | 22
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 2
Arm/Group | Sequence 1: Apremilast Fasted / Fed | Sequence 2: Apremilast Fed / Fasted
Started | 23 | 22
Completed | 22 | 22
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Apremilast: Participants received one dose of 30 mg apremilast administered under fasted conditions and one dose of 30 mg apremilast after a full fat meal.
Arm/Group | Apremilast
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31
  Black or African American | 13
  Asian | 1
  American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Apremilast
Description: Plasma concentrations of apremilast were determined by using a validated liquid chromatography-tandem mass spectrometry assay.
Time Frame: Day 1 of each treatment period at pre-dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The pharmacokinetic (PK) population included all participants who received at least 1 dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Apremilast - Fasted: Participants received a single 30 mg apremilast tablet administered under fasted conditions.
- Apremilast - Fed: Participants received a single 30 mg apremilast tablet administered after a high fat meal.
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 44
ng/mL | 339.86 (26.5) | 333.85 (30.0)
Statistical Analysis 1: Comparison: Apremilast - Fasted vs Apremilast - Fed; To assess the food effect, an analysis of variance model (ANOVA) with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed Cmax of apremilast; Test type: Other — Food was considered to have no effect on the PK of apremilast if the 90% confidence interval (CI) of the geometric least squares (LS) mean ratios for AUC0-t and Cmax were completely contained within the range of 80% to 125%; Ratio of Geometric Least Squares Means = 98.3, 90% CI 2-sided [90.7 to 106.6] — Ratio of the geometric LS means (Fed/Fasted), reported as percentages

2. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was any noxious, unintended, or untoward medical occurrence that appeared or worsened in a participant during the course of this study. It could have been a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE.
Time Frame: From first dose of study drug in Period 1 up to 5 to 10 days after dosing in Period 2, approximately 20 days.
Population: The safety population included all participants who received at least 1 dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 46
Participants
  Any adverse event | 9 | 5
  Adverse events related to study drug | 4 | 3
  Serious adverse events | 0 | 0
  Discontinued due to adverse event | 0 | 2
  Discontinued due to adverse event related to study drug | 0 | 1

3. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Apremilast
Description: as for outcome 1
Time Frame: Day 1 of each treatment period at pre-dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received at least 1 dose of apremilast and had evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 44
hours | 2.50 [0.62 to 5.02] | 3.00 [1.00 to 8.00]
Statistical Analysis 1: Comparison: Apremilast - Fasted vs Apremilast - Fed; Tmax was analyzed by nonparametric methods. The median difference and 90% CI of the median difference were calculated from the Hodges-Lehrmann estimate; Test type: Other; p = 0.0077, Wilcoxon signed-rank test; Median Difference = 0.75, 90% CI 2-sided [0.25 to 1.25] — Median difference (Fed - Fasted) calculated from the Hodges-Lehmann estimate

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) of Apremilast
Description: Plasma concentrations of apremilast were determined by using a validated liquid chromatography-tandem mass spectrometry assay.
  AUC0-t was calculated using the linear trapezoidal method (linear up log down) when concentrations were increasing and the logarithmic trapezoidal method when concentrations were decreasing.
Time Frame: Day 1 of each treatment period at pre-dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received at least 1 dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 44
ng*hr/mL | 3083.05 (34.0) | 3436.39 (33.0)
Statistical Analysis 1: Comparison: Apremilast - Fasted vs Apremilast - Fed; To assess the food effect, an analysis of variance model (ANOVA) with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-t of apremilast; Test type: Other — Food was considered to have no effect on the PK of apremilast if the 90% CI of the geometric LS mean ratios for AUC0-t and Cmax were completely contained within the range of 80% to 125%; Ratio of Geometric LS Means = 112.4, 90% CI 2-sided [109.3 to 115.6] — Ratio of the geometric LS means (Fed/Fasted), reported as percentages

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast
Description: as for outcome 1
Time Frame: Day 1 of each treatment period at pre-dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received at least 1 dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 44
ng*hr/mL | 3157.96 (34.6) | 3506.19 (33.9)
Statistical Analysis 1: Comparison: Apremilast - Fasted vs Apremilast - Fed; To assess the food effect, an ANOVA with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-∞ of apremilast; Test type: Other; Ratio of Geometric Least Squares Means = 112.0, 90% CI 2-sided [108.9 to 115.1] — Ratio of the geometric LS means (Fed/Fasted), reported as percentages

6. Primary Outcome: Estimate of Terminal Elimination Half-life of Apremilast in Plasma (t1/2)
Description: as for outcome 1
Time Frame: Day 1 of each treatment period at pre-dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received at least 1 dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 44
hours | 8.88 (21.2) | 7.99 (18.9)

7. Primary Outcome: Apparent Total Plasma Clearance When Dosed Orally (CL/F) of Apremilast
Description: as for outcome 1
Time Frame: Day 1 of each treatment period at pre-dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received at least 1 dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 44
mL/hr | 9499.80 (34.6) | 8556.28 (33.9)

8. Primary Outcome: Apparent Total Volume of Distribution When Dosed Orally (Vz/F) of Apremilast
Description: as for outcome 1
Time Frame: Day 1 of each treatment period at pre-dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received at least 1 dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Apremilast - Fasted | Apremilast - Fed
Number analyzed (Participants) | 45 | 44
mL | 121735.96 (38.2) | 98582.15 (28.0)

ADVERSE EVENTS:
Time Frame: From first dose of study drug in Period 1 up to 5 to 10 days after dosing in Period 2, approximately 20 days.
Description: Adverse events are reported for all participants who received at least 1 dose of study drug.
Groups:
- Total: Participants received one dose of 30 mg apremilast administered under fasted conditions and one dose of 30 mg apremilast after a full fat meal.
Arm/Group | Apremilast - Fasted | Apremilast - Fed | Total
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 5/45 | 3/46 | 7/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast - Fasted (N=45) | Apremilast - Fed (N=46) | Total (N=46)
Nausea (Gastrointestinal disorders) | 3 | 2 | 5
Headache (Nervous system disorders) | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.